CLINICAL TRIAL: NCT02393807
Title: A Phase 1 Single-dose Open Label 3-way Crossover Study To Evaluate The Bioavailability Of A Spray Dried Dispersion Solid Dose Formulation Of Pf-06260414 Relative To A Suspension Formulation Under Fasted Conditions And The Effect Of Food On The Bioavailability Of The Pf-06260414 Spray Dried Dispersion Solid Formulation In Healthy Subjects
Brief Title: The Bioavailability of a Spray Dried Dispersion Solid Dose Formulation of PF-06260414 Relative to a Suspension Formulation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7411002; SARM FOOD EFFECT & BE (Other: Alias Study Number); SARM FOOD EFFECT &BE (Other: Alias Study Number)
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label single dose crossover study of PF-06260414 (Experimental): This will be a Phase 1, open label, randomized, single dose, 3 period, 3 way crossover study to evaluate the relative bioavailability of solid dose formulation of PF 06260414 under fasted conditions compared to the nanosuspension under fasted conditions
  Interventions: Drug: PF 06260414 solid dose formulation; Drug: PF-06260414 nanosuspension

INTERVENTIONS:
Drug: PF 06260414 solid dose formulation — Single dose of 30 mg PF-06260414 given under fed/fasted conditions
Drug: PF-06260414 nanosuspension — Single dose of 30 mg PF-06260414 given under fasted conditions

SUMMARY:
The current study will investigate the relative bioavailability of a spray dried dispersion solid dose formulation of PF 06260414 administered as a single oral dose of 30 mg of PF 06260414 relative to a single oral dose of 30 mg of PF 06260414 administered as a nanosuspension under fasted or fed conditions in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any condition possibly affecting drug absorption (eg, gastrectomy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Single dose pharmacokinetics under fasted condition: Cmax of PF- 06260414 formulations | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Single dose pharmacokinetics under fasted condition: AUClast of PF- 06260414 formulations | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Single dose pharmacokinetics under fed condition: Cmax of PF- 06260414 formulations | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Single dose pharmacokinetics under fed condition: AUClast of PF- 06260414 formulations | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose

SECONDARY OUTCOMES:
AUCinf of PF-06260414 | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
t½ of PF-06260414 | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
Tmax of PF-06260414 | Hour 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States